CLINICAL TRIAL: NCT01789957
Title: An Open-Label Extension Study of Protocol 2993-112 to Examine the Long-Term Effect on Glucose Control (HbA1c) and Safety and Tolerability of AC2993 Given Two Times a Day to Subjects Treated With Metformin Alone
Brief Title: Extension Study for 2993-112
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2993-112E
Record Dates: First submitted 2013-02-11; First posted 2013-02-12 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label AC2993 (Experimental)
  Interventions: Drug: AC2993

INTERVENTIONS:
Drug: AC2993 — 4-Week transition of AC2993 5 mcg subcutaneously injected twice daily followed by an open-ended period through study termination (up to 52 weeks) of AC2993 10 mcg subcutaneously injected twice daily
  Other Names: Exenatide

SUMMARY:
This multicenter, open-label extension study of Protocol 2993-112 is designed to assess long-term glucose control as measured by HbA1c (glycosylated hemoglobin) and to evaluate long-term safety and tolerability in subjects treated with metformin who receive subcutaneously injected AC2993 (10 mcg) administered twice daily. Subjects completing Protocol 2993-112 are eligible to enroll.

ELIGIBILITY:
All of the following criteria are to be fulfilled for inclusion of an individual in the study unless the sponsor grants an exception:

* Has completed the 30-week triple-blind treatment initiation/active treatment periods in Protocol 2993-112, including all procedures required at the study termination visit (Week 30).
* Male or female. Female individuals must be either 1) postmenopausal as documented by serum FSH measurement unless using estrogen for hormone replacement therapy; or 2) of childbearing potential and used appropriate contraceptive methods (surgical sterility or oral, injected, barrier, intrauterine, or implanted contraceptives) for the duration of Protocol 2993-112. This individual must have a current, negative pregnancy test (human chorionic gonadotropin [HCG], beta subunit) regardless of birth control method used. The individual agrees to continue using birth control throughout the study to prevent pregnancy.
* Able to understand and sign a Protocol 2993-112E-specific informed consent form, communicate with the investigator, and understand and comply with the protocol requirements.

Individuals meeting any of the following criteria are to be excluded from the study unless the sponsor grants an exception:

* Has not completed Protocol 2993-112.
* Female individuals who are pregnant, lactating, or planning to become pregnant.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2002-09; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from Day 1 of Protocol 2993-112 to Week 52 (or termination) | Day 1 of study 2993-112 through extension study termination (up to Week 52)
  Change in HbA1c from Visit 3 (Day 1) of Protocol 2993-112 to Visit 6E (Week 52) of the extension study and to each intermediate visit in the extension study will be calculated and summarized descriptively.
Change in body weight from Day 1 of Protocol 2993-112 to Week 52 (or termination) | Day 1 of study 2993-112 through extension study termination (up to Week 52)
  Change in body weight (KG) from Visit 3 (Day 1) of Protocol 2993-112 to Visit 6E (Week 52) of the extension study and to each intermediate visit in the extension study will be calculated and summarized descriptively.

CONTACTS AND LOCATIONS:
Locations (226):
- United States (219):
  - Pinnacle Research Group, Anniston, Alabama
  - Parkway Medical Center, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Eclectic Family Care, Eclectic, Alabama
  - Winston Physician Services, Haleyville, Alabama
  - Simon Williamson Clinic, Hueytown, Alabama
  - Extended Arm Physicians/ Southern Drug, Montgomery, Alabama
  - Southern Drug Research Network, Tallassee, Alabama
  - Mesa Center for Clinical Research, Chandler, Arizona
  - Clinic of Physicians and Surgeons, Ltd., Mesa, Arizona
  - ANA Ventures, LLC, Mesa, Arizona
  - Lovelace Scientific Resources, Phoenix, Arizona
  - Physicians at the Peak, Phoenix, Arizona
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - First Care Family Doctors, Fayetteville, Arkansas
  - CAVHS, Little Rock, Arkansas
  - Physicians Group Research Clinic, LLC, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Endocrine Metabolic Medical Center, Atherton, California
  - Mitchell Research Group, Inc., Bakersfield, California
  - William Zigrang, M.D., Burlingame, California
  - International Clinical Research Network, Chula Vista, California
  - Arrowhead Regional Medical Center, Colton, California
  - East Bay Clinical Trial Center, Concord, California
  - Medical Group of Encino, Encino, California
  - Mowry Clinical Research, Fremont, California
  - SARC Research Center, Fresno, California
  - Valley Research, Fresno, California
  - Irvine Clinical Research Center, Irvine, California
  - Whittier Institute for Diabetes, La Jolla, California
  - Harriman Jones Medical Group, Long Beach, California
  - Richard Cherlin, M.D., Los Gatos, California
  - Tushar Modi, M.D., Modesto, California
  - Dr. Martinez Medical Clinic, Moreno Valley, California
  - Arroyo Seco Medical Group, Pasadena, California
  - Elke Jost-Vu, M.D., Rancho Mirage, California
  - Comprehensive Diabetes-Endocrine Medical Associates, Redwood City, California
  - nTouch, San Diego, California
  - Radiant Research, San Diego, California
  - San Diego Endocrine and Medical Clinic, San Diego, California
  - Veterans Medical Research Foundation, San Diego, California
  - Diabetes Research Institute of Mills Peninsula, San Mateo, California
  - Advanced Clinical Research Institute, Santa Ana, California
  - Pacific Clinical Research, Santa Monica, California
  - West Coast Clinical Trials, Signal Hill, California
  - Protocare Trials at Sharp Mission Park, Vista, California
  - Diablo Clinical Research, Walnut Creek, California
  - University of Colorado-Barbara Davis Center for Childhood Diabetes, Denver, Colorado
  - Pheonix International Medicine Associates, Waterbury, Connecticut
  - Health Core at Health Care Center Christiana, Newark, Delaware
  - Medstar Clinical Research, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - Morton Plant Mease Health Care, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Atlantic Institute of Clinical Research, Daytona Beach, Florida
  - Halifax Clinical Research Institute, Daytona Beach, Florida
  - Internal Medical Associates, Fort Myers, Florida
  - Clin Sci International, Gainesville, Florida
  - University of FL, Gainesville, Florida
  - South Florida Clinical Research Center, Hollywood, Florida
  - Health Trials 3000, Jacksonville, Florida
  - Jupiter Research Institute, Jupiter, Florida
  - ICSL Clinical Studies, Maitland, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - VRG Research, Orlando, Florida
  - Highland Lakes Medical Center, Palm Harbor, Florida
  - Tallahassee Endocrine Associates, Tallahassee, Florida
  - Biostator / USF Diabetes Center, Tampa, Florida
  - Tampa Medical Group, Tampa, Florida
  - Diabetes and Endocrine Associates of the Treasure Co, Vero Beach, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Radiant Research, West Palm Beach, Florida
  - ICSL-Clinical Studies, Atlanta, Georgia
  - Clinical Research Atlanta, Atlanta, Georgia
  - Columbus Metabolic Foundation, Columbus, Georgia
  - nTouch Research Corporation, Decatur, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Radiant Research, Honolulu, Hawaii
  - St. Luke's Family Health, Meridian, Idaho
  - University Primary Care Center at Belvidere, Belvidere, Illinois
  - Northwestern Memorail Physicians Group, Chicago, Illinois
  - Illinois Center for Clinical Trials, Chicago, Illinois
  - Cook County Hospital, Chicago, Illinois
  - Lake Forest Internal Medicine, Libertyville, Illinois
  - Winchester Research Group, Libertyville, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Diabetes and Endocrinology, Springfield, Illinois
  - Medical Group of Fort Wayne, Fort Wayne, Indiana
  - Indiana University Outpatient Clinical Research, Indianapolis, Indiana
  - American Health Network, Indianapolis, Indiana
  - Center for Metabolic and Hormonal Disorders, Indianapolis, Indiana
  - nTouch Research Corporation, South Bend, Indiana
  - Ramona Holiday Diabetes Center, Des Moines, Iowa
  - Diabetes Clinical Research and Programs, Iowa City, Iowa
  - Lipid, Atherosclerosis & Metabolic Clinic, Kansas City, Kansas
  - Kentucky Diabetes Center, Lexington, Kentucky
  - Central Kentucky Research Associates, Lexington, Kentucky
  - University of Kentucky Metabolic Research Group, Lexington, Kentucky
  - MedResearch, Inc., Louisville, Kentucky
  - Drug Research Services, Metairie, Louisiana
  - New Orleans Institute of Clinical Investigation, New Orleans, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Diabetes, Endocrine and Nutrition Center, Bangor, Maine
  - VA Medical Center, Baltimore, Maryland
  - St. Agnes Health Care, Baltimore, Maryland
  - Doctors Research Associates of Maryland, Lanham, Maryland
  - University of Michigan-Endocrinology and Metabolism, Ann Arbor, Michigan
  - Grunberger Diabetes Medical Center, Bloomfield Hills, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Grand Rapids Associated Interns, Grand Rapids, Michigan
  - Westside Family Medical Center, Kalamazoo, Michigan
  - Mayo Clinic, Division of Endocrinology and Metabolism, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Diabetes and Endocrinology Specialists, Chesterfield, Missouri
  - Midwest Pharmaceutical Research, City of Saint Peters, Missouri
  - Medical Arts Research Collaborative, Excelsior Springs, Missouri
  - St Lukes Lipid and Diabetes Research Center, Kansas City, Missouri
  - Mid Missouri Research Specialists, Inc., Rolla, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Radiant Research, St Louis, Missouri
  - Mercury Street Medical, Butte, Montana
  - Creighton Diabetes Center, Omaha, Nebraska
  - Lovelace Scientific Resources, Las Vegas, Nevada
  - ICSL, Las Vegas, Nevada
  - Endocrinology and Diabetes Consultants, P.C., Dover, New Hampshire
  - HIS Clinical Research, Jersey City, New Jersey
  - Radiant Research, Moorestown, New Jersey
  - Matrix Research Institute, Mount Laurel, New Jersey
  - New Jersey Physicians, Passaic, New Jersey
  - Anderson and Collins Clinical Research, Inc., South Plainfield, New Jersey
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - SUNY Downstate, Brooklyn, New York
  - Medical Network Services, P.C., Brooklyn, New York
  - Winthrop University Hospital, Mineola, New York
  - St. Lukes Roosevelt Hospital, New York, New York
  - Irving Diabetes Research Unit at Columbia University, New York, New York
  - Naomi Berrie Diabetes Center at Columbia University, New York, New York
  - Heights Medical Care, New York, New York
  - Rochester Clinical Research, Rochester, New York
  - Albert Einstein College of Medicine of Yeshiva University, The Bronx, New York
  - DOCS at Beth Israel Medical Center, Yonkers, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Charlotte Clinical Research, Charlotte, North Carolina
  - UNC Diabetes Care Center, Durham, North Carolina
  - Unifour Medical Research, Hickory, North Carolina
  - New Hanover Medical Research Associates, Wilmington, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Rapid Medical Research, Cleveland, Ohio
  - Ohio State University-Division of Endocrinology, Columbus, Ohio
  - Radiant Research, Columbus, Ohio
  - University Mednet, Mentor, Ohio
  - Comprehensive Research Services, Inc., Mogadore, Ohio
  - North Coast Institute of Diabetes and Endocrinology, Westlake, Ohio
  - Prime Care Clinical Research, Clinton, Oklahoma
  - COR Clinical Research, Oklahoma City, Oklahoma
  - OU Health Sciences Center, Oklahoma City, Oklahoma
  - nTouch Research Corporation, Oklahoma City, Oklahoma
  - Utica Park Clinic, Tulsa, Oklahoma
  - Americas Doctors, Medford, Oregon
  - Medford Medical Clinic, Medford, Oregon
  - Radiant Research, Portland, Oregon
  - Portland Diabetes and Endocrinology Center, Portland, Oregon
  - Pacific Coast Clinical Coordinators, Inc., Portland, Oregon
  - Legacy Clinical Research, Portland, Oregon
  - Physicians for Clinical Research, Camp Hill, Pennsylvania
  - Argus Research Laboratories, Horsham, Pennsylvania
  - Thomas Jefferson University Diabetes Research Center, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Philadelphia Health Associates, Philadelphia, Pennsylvania
  - Elite Medical Research, Inc., Sellersville, Pennsylvania
  - Tipton Medical and Diagnostic Center, Tipton, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - ICSL-Providence, East Providence, Rhode Island
  - Radiant Research, Charleston, South Carolina
  - CNS Clinical Trials, Chester, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Tennessee Valley Clinical Research Associates, Alcoa, Tennessee
  - Integrity Clinical Research, Jackson, Tennessee
  - Harmony Clinical Research, Johnson City, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Endocrine Consultants of ET, Knoxville, Tennessee
  - The Endocrine Clinic, Memphis, Tennessee
  - Integrity Clinical Research, Milan, Tennessee
  - Mid State Endocrine Associates, Nashville, Tennessee
  - Israel A. Hartman, M.D., Arlington, Texas
  - Central Texas Clinical Research, Austin, Texas
  - Dallas Diabetes and Endocrinology Research Center, Dallas, Texas
  - Rafael Canadas M.D., P.A., Dallas, Texas
  - Texas Tech University Health Sciences-Internal Medicine, El Paso, Texas
  - Internal Medicine Associates, El Paso, Texas
  - Lanier Education Research Network, Fort Worth, Texas
  - North Texas Clinical Research, Irving, Texas
  - Dr. Humberto Bruschetta, Kingsville, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - South Texas Applied Research, McAllen, Texas
  - Sun Research Institute, San Antonio, Texas
  - University of Texas Health Sciences Center-Texas Diabetes Institute, San Antonio, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - SAM Clinical Research, San Antonio, Texas
  - Utah Diabetes Center at the University of Utah, Salt Lake City, Utah
  - Salt Lake Research, Salt Lake City, Utah
  - Medical Associates of Northern Virginia, Arlington, Virginia
  - Clinical Research Center-Eastern Virginia Medical School, Norfolk, Virginia
  - Drs. Wigand, Wasserman, and Associates, Richmond, Virginia
  - Evergreen Diabetes & Endocrinology, Kirkland, Washington
  - Olympic Medical Services, Lacey, Washington
  - West Olympia Internal Medicine, Olympia, Washington
  - Rainier Clinical Research Center, Renton, Washington
  - Northside Internal Medicine, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Julia M. Hutchinson, M.D., Spokane, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - Hyperion Clinical Research, Charleston, West Virginia
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - University of Wisconsin West Clinic, Madison, Wisconsin
  - Midwest Endocrinology Associates, Milwaukee, Wisconsin
  - VRG Research, Milwaukee, Wisconsin
- Canada (7):
  - Calgary Metabolic Education and Research Center, Calgary, Alberta
  - Walter McKenzie Health Sciences Centre, Edmonton, Alberta
  - St. Paul's Hospital, Research Services, Vancouver, British Columbia
  - Health Sciences Center, Winnipeg, Manitoba
  - University of Western Ontario, London, Ontario
  - McGill Nutrition and Food Science Center, Montreal, Quebec
  - Centre Hospitalier, Ste. Foy, Quebec